CLINICAL TRIAL: NCT03610451
Title: Influence of Floatation-REST (Reduced Environmental Stimulation Therapy) on Anorexia Nervosa
Brief Title: Floatation-REST and Anorexia Nervosa
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Laureate Institute for Brain Research, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-001-02
Record Dates: First submitted 2018-03-19; First posted 2018-08-01 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Anorexia Nervosa
Keywords: Anorexia nervosa; Floatation therapy
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Intervention Model Description: Pragmatic randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Floatation-REST (Experimental): Participants will float supine in a pool of water saturated with epsom salt, in a light and sound attenuated chamber, for up to 60 minutes, on 8 separate occasions. Ratings of the experience will be collected before and after each float.
  Interventions: Behavioral: Floatation-REST plus usual care
- Usual care (Other): Participants will be assessed along the same time periods, i.e., before and after a 60 minute window, on 8 separate occasions. Ratings of the experience will be collected before and after each time period.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Floatation-REST plus usual care — Individuals will receive Floatation-REST plus usual care. Floating creates an environment with minimal visual, auditory, tactile, proprioceptive, and thermal input to the brain. The float rooms are lightproof and soundproof. A high concentration Epsom salt water solution allows individuals to effortlessly float on their back while remaining completely still, reducing both proprioceptive and tactile input to the brain. The temperature of the water is calibrated to the temperature of the skin (~94° F) and the temperature of the air is calibrated to the temperature of the water, making it difficult to discern the boundary between air and water, thus reducing thermal input to the brain while minimizing the need for thermoregulation of the skin.
  Arms: Floatation-REST
Behavioral: Usual care — Individuals will receive usual care on the inpatient unit of the Laureate Eating Disorders Program.
  Arms: Usual care

SUMMARY:
The study proposed in this protocol aims to document the effect of Floatation-REST (reduced environmental stimulation therapy) on symptoms of anorexia nervosa.

DETAILED DESCRIPTION:
Flotation-REST (reduced environmental stimulation therapy) alters the balance of sensory input by systematically attenuating signals from the visual, auditory, thermal, tactile, vestibular, and proprioceptive systems. Previous research has shown that this heightens interoceptive awareness and reduces anxiety in clinically anxious populations. Anorexia nervosa (AN) is characterized by elevated anxiety, distorted body image, and disrupted interoception, raising the question of whether floatation therapy might positively impact these symptoms. A recent safety study found that Floatation-REST was well tolerated by individuals weight-restored outpatients with current or prior AN. Additionally, participants reported improvements in affective state and body image disturbance following floating, raising the possibility that this intervention might be investigated for clinical benefit in more acutely ill cases.

The primary aim of this study is to begin to examine the effect of Floatation-REST on body image disturbance in inpatients with AN. Secondary aims including determining whether Floatation-REST has an impact on anxiety, emotional distress, eating disorder severity, functional ability, and interoception.

ELIGIBILITY:
Inclusion Criteria:

* Primary clinical diagnosis of anorexia nervosa
* Receiving inpatient treatment for eating disorder
* Body mass index greater than or equal to 16
* No new medication prescription in the week prior to study randomization
* Independently ambulatory
* No current evidence of orthostatic hypotension
* Ability to lay flat comfortably
* Possession of a smartphone with data plan
* English proficiency

Exclusion Criteria:

* Active suicidal ideation
* Active cutting or skin lacerating behaviors
* Orthostatic hypotension (defined as a drop of ≥ 20 mm Hg in systolic BP or a drop of ≥ 10 mm Hg in diastolic BP when measured shortly after transitioning from lying down to standing)
* Comorbid schizophrenia spectrum or other psychotic disorder

Ages: 13 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 68 (Actual)
Dates: Start 2018-03-16 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Body image dissatisfaction score on the Photographic Figure Rating Scale | Through study completion, an average of 1 year
  Average of the absolute change in body image dissatisfaction from pre to post float across all eight floats (score range: 0 to 10; larger changes indicate greater severity of body image dissatisfaction)

SECONDARY OUTCOMES:
Anxiety on the Spielberger State Trait Anxiety Inventory | Through study completion, an average of 1 year
  Average of the change in anxiety rating from pre to post float across all eight float (range 20 to 80, higher scores indicate greater severity of anxiety)
Anxiety on the NIH Promis Anxiety Scale | Through study completion, an average of 1 year
  Average of the change in anxiety rating from pre to post float across all eight float (range 6 to 30, higher scores indicate greater severity of anxiety)
Anxiety sensitivity on the Anxiety Sensitivity Index-3R | Through study completion, an average of 1 year
  Change in anxiety sensitivity after the final float relative to baseline (range 0 to 96, higher scores indicate greater severity of anxiety sensitivity)
Eating disorder severity on the Eating Disorder Examination Questionnaire | Through study completion, an average of 1 year
  Change in eating disorder severity after the final float relative to baseline (range 0 to 6, larger scores indicate greater severity of eating disorder)
Functional ability on the Sheehan Disability Questionnaire | Through study completion, an average of 1 year
  Change in functional ability after the final float relative to baseline (range 0 to 30, higher scores indicate greater severity of disability)
Body image disturbance on the Body Image States Scale | Through study completion, an average of 1 year
  Change in body image disturbance after the final float relative to baseline (range 0 to 48, higher scores indicate greater severity of body image disturbance)
Interoceptive self report on the Multidimensional Interoceptive Awareness Scale | Through study completion, an average of 1 year
  Change in total interoceptive awareness score after the final float relative to baseline (range 0 to 160, higher scores indicating greater interoceptive awareness)
Body image disturbance on the Body Appreciation Scale-2 | Through study completion, an average of 1 year
  Change in body image disturbance score after the final float relative to baseline (range 10 to 50, higher scores indicating reduced severity of body image disturbance)

CONTACTS AND LOCATIONS:
Overall Officials: Sahib Khalsa, MD, PhD, Principal Investigator — Laureate Institute for Brain Research
Locations (1):
- Laureate Institute for Brain Research, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Choquette EM, Flux MC, Moseman SE, Chappelle S, Naegele J, Upshaw V, Morton A, Paulus MP, Feinstein JS, Khalsa SS. The impact of floatation therapy on body image and anxiety in anorexia nervosa: a randomised clinical efficacy trial. EClinicalMedicine. 2023 Aug 29;64:102173. doi: 10.1016/j.eclinm.2023.102173. eCollection 2023 Oct. PMID 37936658